CLINICAL TRIAL: NCT05206019
Title: Study to Evaluate Pharmacokinetic and Safety of Albuvirtide Between Intravenous Drip and Intravenous Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Frontier Biotechnologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FB-ABWT-402
Record Dates: First submitted 2021-12-30; First posted 2022-01-25 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — albuvirtide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- cohort 1: Albuvirtide (Experimental): Single dose of 320 mg by intervenous drop infusion for 45 min
  Interventions: Drug: Albuvirtide
- cohort 2: Albuvirtide (Experimental): Single dose of 320 mg by intervenous injection for 0.5 min
  Interventions: Drug: Albuvirtide
- cohort 3: Albuvirtide (Experimental): Single dose of 320 mg by intervenous injection for 3 min
  Interventions: Drug: Albuvirtide

INTERVENTIONS:
Drug: Albuvirtide — Long-Acting HIV-1 Fusion Inhibitor (chemically modified peptide targeting HIV-1 gp41)

SUMMARY:
This is a single-center,randomized,open, single-dose, parallel-design study, which will be only enrolled Chinese healthy volunteers.

DETAILED DESCRIPTION:
30 Chinese volunteers will be enrolled to assess the pharmacokinetic and safety of Albuvirtide in two different Administration methods. All subjects are required to collect PK blood samples before and after administration.

30 healthy subjects will be randomized into three cohorts ( cohorts A, B and C) in 1:1:1 ratio, with 10 subjects in each cohort. The subjects will receive a single dose of 320 mg of albuvirtide by iv infusion for 45 min or by iv bolus for 0.5 min or 3 min, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18-55, healthy volunteers (including the threshold, based on time of signing informed consent form).
2. BMI of 19 to 26 kg/m2 (including the threshold), with male ≥ 50 kg and female ≥ 45 kg.
3. Subjects and their partners agreed never to have children from 2 weeks prior to screening until 6 months after administration and volunteered to use effective contraception, regardless of sperm or oocyte donation plans.

Exclusion Criteria:

1. Allergic to investigational drug or allergic constitution .
2. With difficulty in intravenous administration/blood collection or a history of dizziness from needles and blood.
3. Have substance abuse in the past 5 years or used drugs in the past 3 months prior to screening, or drug tested positive.
4. Smoked an average of >5 cigarettes per day in the 3 months prior to screening or were unable to stop using any tobacco-based products during the study.
5. Consumption of an average of >14 units of alcohol per week (1 unit of alcohol ≈ 360 mL of beer or 45 mL of spirits with 40% alcohol content or 150 mL of wine) in the past 3 months prior to screening, or inability to abstain from alcohol during the trial, or positive blood test for alcohol
6. Any drugs that inhibit or induce hepatic CYP3A metabolizing enzymes (e.g., inducers - barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; inhibitors - ketoconazole, itraconazole, cimetidine, diltiazem, macrolides, nitroimidazoles, sedative-hypnotics, verapamil, fluoroquinolones, antihistamines) within 30 days prior to screening.
7. Any use of prescription, over-the-counter or herbal medicines and supplements within 14 days prior to screening
8. Received vaccination within 4 weeks prior to screening or planned vaccination during the study.
9. Consumption of dragon fruit, mango, grapefruit, carambola or food or drink prepared from them within 48 hours prior to admission.
10. Have special requirements for diet.
11. History or presence of any disease or condition which might compromise the Neurological, cardiovascular, hematological, hepatic, renal, gastrointestinal, respiratory, metabolic, endocrine, immune, and skeletal systems or any other body system.
12. During the screening period, vital signs, physical examination, laboratory tests,12-lead electrocardiogram or chest radiograph is abnormal with clinically significant.
13. During the screening period, virological testing, hepatitis B surface antigen or e antigen, hepatitis C antibody, syphilis spirochete antibody, or human immunodeficiency virus (HIV) antibody is positive.
14. Women who tested positive for pregnancy at screening or baseline or lactating
15. Participated in other drug clinical trials and took medication within 3 months prior to screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2022-04-17 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Area under curve | Day 0-Day 57
  The area under the plase of the last measurable The area under the curve of the last measurable concentration (AUCt)
Peak concentration | Day 0-Day 57
  Maximum observed plasma concentration (Cmax)
Peak time | Day 0-Day 57
  Time to Cmax ( Tmax)
half-time | Day 0-Day 57
  Time for blood concentration to drop by half-time（t1/2）

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Day 0-Day 63
  Incidence of Treatment-Emergent Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Anhui Medical University, Hefei, China